CLINICAL TRIAL: NCT04759833
Title: Phase 3, Multicenter, Randomized Study With 2 Different Doses of Prucalopride Administered to Male and Female Pediatric Subjects Aged 6 Months to 17 Years With Functional Constipation, Consisting of a 12-week Double-blind, Placebo-controlled Part (Part A) to Evaluate Efficacy and Safety Followed by a 36-week Double-blind Extension Part (Part B) to Document Long-term Safety up to Week 48
Brief Title: A Study of Prucalopride For Functional Constipation in Children and Teenagers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Data Monitoring Committee (DMC) decision; terminated due to futility, with no safety concerns; FDA agreement to terminate the study.
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-555-3010; 2022-003221-22 (EudraCT Number)
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Placebo (Placebo Comparator): Participants weighing <50 kilograms (kg) will draw equal volumes from two bottles of placebo oral solution to account for the daily dose assigned or participants weighing ≥ 50 kg will receive two placebo oral tablets, once daily (QD), during 12 weeks in Part A. Prucalopride matching placebo (oral solution or tablet) will be dosed depending on the participant's body weight (BW) at the randomization visit.
  Interventions: Other: Placebo
- Part A: Low Dose Prucalopride (Experimental): Participants weighing <50 kg will receive 0.04 milligrams per kilogram (mg/kg) of prucalopride oral solution (will draw the required volume from one bottle of 0.4 milligram per milliliter [mg/mL] and one bottle of placebo oral solution), QD or participants weighing ≥50 kg will receive one 2 milligram (mg) of prucalopride oral tablet and one placebo oral tablet, QD, during 12 weeks in Part A. Prucalopride (oral solution or tablet) will be dosed depending on the participant's BW at the randomization visit.
  Interventions: Drug: Prucalopride
- Part A: High Dose Prucalopride (Experimental): Participants weighing <50 kg will receive 0.08 mg/kg of prucalopride oral solution (will draw the required volume from two bottles of 0.4 mg/mL to account for the daily dose assigned), QD or participants weighing ≥50 kg will receive two 2 mg of prucalopride oral tablets, QD, during 12 weeks of treatment period in Part A. Prucalopride (oral solution or tablet) will be dosed depending on the participant's BW at the randomization visit.
  Interventions: Drug: Prucalopride
- Part B: Low Dose Prucalopride (Experimental): Participants weighing <50 kg will receive 0.04 mg/kg of prucalopride oral solution (will draw the required volume from one bottle of 0.4 mg/mL and one bottle of placebo oral solution to account for the daily dose assigned), QD or participants weighing ≥50 kg will receive one 2 mg of prucalopride oral tablet and one placebo oral tablet, QD, for 36 weeks during the 40-week Part B Period. Prucalopride (oral solution or tablet) will be dosed depending on the participant's BW at the randomization visit.
  Interventions: Drug: Prucalopride
- Part B: High Dose Prucalopride (Experimental): Participants weighing <50 kg will receive 0.08 mg/kg of prucalopride oral solution (will draw the required volume from two bottles of 0.4 mg/mL to account for the daily dose assigned), QD or participants weighing ≥50 kg will receive two 2 mg of prucalopride oral tablets, QD, for 36 weeks during the 40-week Part B Period. Prucalopride (oral solution or tablet) will be dosed depending on the participant's BW at the randomization visit.
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — Prucalopride oral solution or oral tablets.
  Other Names: TAK-555; Prucalopride succinate
  Arms: Part A: High Dose Prucalopride; Part A: Low Dose Prucalopride; Part B: High Dose Prucalopride; Part B: Low Dose Prucalopride
Other: Placebo — Prucalopride-matching placebo oral solution or oral tablets.
  Arms: Part A: Placebo

SUMMARY:
Functional constipation is a condition when it is very hard to pass a stool that is not due to any other health problem or to medicines being taken. This condition is more common in children and teenagers.

This study has 2 parts:

The main aim of the 1st part of the study is to learn if a medicine called prucalopride can improve bowel movements in children and teenagers with functional constipation. Another aim is to check for side effects from 2 different doses of prucalopride. The main aim of the 2nd part of the study is to continue to check for side effects from 2 different doses of prucalopride.

In the 1st part, at the first visit, the study doctor will check who can take part. Participants who take part will be picked for 1 of 3 treatments by chance.

* A low dose of prucalopride once a day.
* A higher dose of prucalopride once a day.
* A placebo once a day. In this study, a placebo will look like prucalopride but will not have any medicine in it. Participants will be treated with prucalopride or a placebo for 12 weeks.

Participants who took prucalopride will continue to the 2nd part of the study. They will have the same treatment as they did in the 1st part of the study. They will continue with their treatment for another 36 weeks. Participants who took placebo in the 1st part of the study will receive prucalopride in the 2nd part of the study. They will be picked for a low dose or a high dose of prucalopride by chance.

Participants will visit the clinic a few times during treatment. The clinic staff will also telephone the participants, or their parents or caregivers throughout treatment for a check-up 4 weeks after last treatment, the clinic staff will telephone the participants, or their parents or caregivers for a final check-up.

DETAILED DESCRIPTION:
This study consists of a 12-week double-blind, placebo-controlled part (Part A) followed by a 36-week double-blind safety extension part (Part B). Participants aged 3 to 17 years are planned for randomization in a 1:1:1 ratio to the Low Dose Group, High Dose Group, or matching placebo (placebo-controlled part [Part A]). After completion of Part A, participants in the placebo group will be re-randomized in a 1:1 ratio to the Low Dose Group or the High Dose Group (safety extension part [Part B]). Randomization at study entry will be stratified by toilet-trained status.

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or their parent(s)/caregiver(s)/legally authorized representative(s) have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed, and dated (personally or via parent[s]/caregiver[s]/legally authorized representative[s]) informed consent/assent as applicable to participate in the study.

Note: Participants and/or parent(s)/caregiver(s)/legally authorized representative(s) (where appropriate depending on age and local regulation) can also provide consent/assent to the sparse Pharmacokinetic (PK) sampling in this study.

* Toilet-trained participants 3 years to 17 years of age, inclusive, or non-toilet-trained participants 6 months to 17 years of age, inclusive.
* Participant weighs greater than or equal to (>=) 5.5 kilograms (kg) (12 pounds [lbs]).
* Male, or non-pregnant, non-lactating female participants who are sexually active and agree to comply with the applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Note: All female participants >= 12 years and/or female participants lesser than (<) 12 years who have started menarche must have a negative serum pregnancy test at screening.

- Participant meets modified Rome IV criteria:

* For child/adolescent (aged > 4 years) functional constipation (H3a):

Participants must have lesser than or equal to (<=) 2 defecations per week and 1 or more of the following occurring at least once per week for a minimum of 1 month:

* >= 1 episode of fecal incontinence per week (only for participants after the acquisition of toileting skills).
* History of retentive posturing or excessive volitional stool retention.
* History of painful or hard bowel movements (BMs).
* Presence of large fecal mass in rectum.
* History of large diameter stools which can obstruct the toilet. In addition, the participant does not satisfy sufficient criteria for a diagnosis of irritable bowel syndrome (IBS) and, after appropriate evaluation, the participants symptoms cannot be fully explained by another medical condition.

For infants/toddler (aged 6 months to <= 4 years) functional constipation (G7):

Participants must have <= 2 defecations per week and >= 1 month of at least 1 of the following:

* History of excessive stool retention
* History of painful or hard BMs
* History of large-diameter stools (in the diaper)
* Presence of a large fecal mass in the rectum

In toilet-trained children, the following additional criteria may be used:

* At least 1 episode/week of incontinence after the acquisition of toileting skills
* History of large-diameter stools which may obstruct the toilet - Participant and/or parent(s)/caregiver(s)/legally authorized representative(s) is willing to discontinue any laxatives during the screening period up to disimpaction and agrees to adhere to the protocol-specified disimpaction and rescue medication rules, if applicable.

To be evaluated prior to randomization:

* Participant has an average of < 3 SBMs (defecations) per week during the screening period and prior to the disimpaction.
* Participant or legally authorized representative (dependent on participant age) is compliant with completing the electronic diary for at least 7 consecutive days preceding the disimpaction.

Exclusion Criteria:

* Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product (IP), or clinical or laboratory assessments.
* Any clinically significant abnormal findings on the electrocardiogram (ECG) that indicates a dysrhythmia or conduction abnormalities (such as abnormal heart rate, PR, QRS, or QT).
* Major cardiovascular disease such as: cardiomyopathy, cardiac insufficiency, uncorrected congenital heart disease, symptomatic valve disorders, or septal defects.
* Current or relevant history of physical or psychiatric illness (e.g. severe autism, depression, etc.), any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the IP or procedures.
* Non-retentive fecal incontinence.
* Intestinal perforation or obstruction due to structural or functional disorder of the gut wall, obstructive ileus, severe inflammatory conditions of the intestinal tract such as Crohn's disease, ulcerative colitis, and toxic megacolon/megarectum.
* Current use of any medication (including over-the-counter, herbal, or homeopathic preparations) that could affect (improve or worsen) the condition being studied (e.g. opioids), or could affect the action, absorption, or disposition of the IP, or clinical or laboratory assessment. (Current use is defined as use within the past 5 days).
* Participants with renal impairment:

  * Participants <= 2 years of age with serum creatinine greater than normal (screening sample results using central laboratory pediatric reference ranges).
  * Participants > 2 years of age with severe renal impairment or end stage renal disease (estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m^2).
* Known or suspected intolerance or hypersensitivity to the IP(s), closely-related compounds, or any of the stated ingredients.
* Known history of alcohol or other substance abuse within the last year.
* Within 30 days prior to the first dose of the IP in the current study:

  * Have used any IP.
  * Have been enrolled in a clinical study (including vaccine studies) that may or may not include the administration of an IP that, in the investigator's opinion, may impact this study.
* Participant used prucalopride within 10 days prior to the first dose of the IP or has been unsuccessfully treated with prucalopride before.
* Participant meets Rome IV criteria for other Child/Adolescent Functional Gastrointestinal Disorders (FGID) (H1 - H2 and H3b).
* Participant with secondary causes of constipation:

  * Endocrine disorders (e.g., hypopituitarism, hypothyroidism, hypercalcemia, pheochromocytoma, glucagon-producing tumors) unless these are controlled by appropriate medical therapy. Participant with uncontrolled diabetes mellitus is to be excluded
  * Metabolic disorders (e.g. porphyria, uremia, hypokalemia, hypothyroidism, amyloid neuropathy), unless controlled by appropriate medical therapy
  * Neurological disorders (e.g. cerebral tumors, cerebrovascular accidents, multiple sclerosis, meningocele, aganglionosis, hypoganglionosis, hyperganglionosis, autonomic neuropathy, spinal cord injury, Chagas disease
  * Organic disorders (known or suspected) of the large bowel (e.g. obstruction from any cause including biliary obstruction, malignancy, intestinal perforation, obstructive ileus, pseudo-obstruction, history of or current anorectal malformations, severe inflammation of the intestinal tract, such as Crohn's disease, ulcerative colitis or toxic megacolon/megarectum, Hirschsprung's disease)
  * Celiac disease, cow milk allergy
  * Surgery: history of gastrointestinal surgery related or possibly related to the presence of constipation
  * Lactose intolerance
* Any of the following clinically significant abnormalities of serum biochemistry:

  * Serum aspartate aminotransferase (AST) >1.5 times upper limit of normal (ULN) at screening.
  * Serum alanine aminotransferase (ALT) >1.5 times ULN at screening.
  * Total bilirubin outside the age-adjusted normal range, except for participants with Gilbert's syndrome.
* Any significant underlying liver disease.
* Participant is not able to swallow the IP (liquid or tablet).
* Participant is pregnant or planning to get pregnant during study period.

To be evaluated prior to randomization:

* Participant has used other disimpaction medication in lieu of the protocol-provided medication.
* Participant has used non-protocol approved medications to induce BMs during the screening period or disimpaction.
* The participant has failed the disimpaction based on the investigator's assessment.
* Worsening of depression and emergence of suicidal thoughts.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (41):
- United States (41):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Novak Clinical Research, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, Davis Department of Pediatrics, Sacramento, California
  - University of California, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Direct Helpers Research Center, Hialeah, Florida
  - Pediatric & Adult Research Center, Kissimmee, Florida
  - Auzmer Research, Lakeland, Florida
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Orlando Health - APH Center for Digestive Health and Nutrition, Orlando, Florida
  - The University of Chicago Medical Center, Chicago, Illinois
  - GI Pediatric Subspecialty Clinic, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Willis-Knighton Center for Pediatric Gastroenterology & Advanced Endoscopy, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - CUMC Pediatrics-GI, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Cyn3rgy Research & Development, Gresham, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - GI For Kids, Knoxville, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Tekton Research, Inc., Beaumont, Texas
  - Cedar Health Research, Dallas, Texas
  - Allure Health LLC, Friendswood, Texas
  - Texas Children's Hospital, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - Pediatric Center, Richmond, Texas
  - University of Utah, Salt Lake City, Utah
  - Pediatric Specialist of Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Cuffari C, Spalding W, Achenbach H, Thakur M, Gabriel A. Design of a phase 3, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of prucalopride in pediatric patients with functional constipation. Contemp Clin Trials Commun. 2023 Apr 30;33:101144. doi: 10.1016/j.conctc.2023.101144. eCollection 2023 Jun. PMID 37215389
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60363ce520847c001e116bdd

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 42 investigative sites in the United States from 13 July 2021 to 13 November 2023.
Pre-assignment Details: A total of 175 participants with a diagnosis of functional constipation were enrolled and randomized in a 1:1:1 ratio to receive either prucalopride at low dose, high dose, or matching placebo in Part A of the study depending on their body weight. All participants who completed Part A entered Part B, and those in the placebo group of Part A were re-randomized based on their weight in a 1:1 ratio to receive either prucalopride at a low or high dose in Part B of the study.
Groups:
- Part A: Placebo: Participants weighing <50 kilograms (kg) drew equal volumes from two bottles of placebo oral solution to account for the daily dose assigned or participants weighing ≥50 kg received two placebo oral tablets, once daily (QD), during 12 weeks in Part A. Prucalopride matching placebo (oral solution or tablet) were dosed depending on the participant's body weight (BW) at the randomization visit.
- Part A: Low Dose Prucalopride: Participants weighing <50 kg received 0.04 milligrams per kilogram (mg/kg) of prucalopride oral solution (drew the required volume from one bottle of 0.4 milligram per milliliter [mg/mL] and one bottle of placebo oral solution), QD or participants weighing ≥50 kg received one 2 milligram (mg) of prucalopride oral tablet and one placebo oral tablet, QD, during 12 weeks in Part A. Prucalopride (oral solution or tablet) were dosed depending on the participant's BW at the randomization visit.
- Part A: High Dose Prucalopride: Participants weighing <50 kg received 0.08 mg/kg of prucalopride oral solution (drew the required volume from two bottles of 0.4 mg/mL to account for the daily dose assigned), QD or participants weighing ≥50 kg received two 2 mg of prucalopride oral tablets, QD, during 12 weeks of treatment period in Part A. Prucalopride (oral solution or tablet) were dosed depending on the participant's BW at the randomization visit.
- Part B: Low Dose Prucalopride: Participants weighing <50 kg received 0.04 mg/kg of prucalopride oral solution (drew the required volume from one bottle of 0.4 mg/mL and one bottle of placebo oral solution to account for the daily dose assigned), QD or participants weighing ≥50 kg received one 2 mg of prucalopride oral tablet and one placebo oral tablet, QD, for 36 weeks during the 40-week Part B Period. Prucalopride (oral solution or tablet) were dosed depending on the participant's BW at the randomization visit.
- Part B: High Dose Prucalopride: Participants weighing <50 kg received 0.08 mg/kg of prucalopride oral solution (drew the required volume from two bottles of 0.4 mg/mL to account for the daily dose assigned), QD or participants weighing ≥50 kg received two 2 mg of prucalopride oral tablets, QD, for 36 weeks during the 40-week Part B Period. Prucalopride (oral solution or tablet) were dosed depending on the participant's BW at the randomization visit.
Period: PartA:Placebo-controlled Period(12Weeks)
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
Started | 56 | 60 | 59 | 0 | 0
Completed | 46 | 49 | 39 | 0 | 0
Not Completed | 10 | 11 | 20 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 4 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 2 | 3 | 0 | 0
Not completed — Withdrawal of Consent by Participant | 5 | 3 | 9 | 0 | 0
Not completed — Noncompliance with Study Drug | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Period: Part B:Safety Extension Period(40 Weeks)
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
Started | 0 | 0 | 0 | 72 | 62
Completed | 0 | 0 | 0 | 37 | 28
Not Completed | 0 | 0 | 0 | 35 | 34
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 21 | 16
Not completed — Withdrawal of Consent by Participant | 0 | 0 | 0 | 4 | 8
Not completed — Reason not Specified | 0 | 0 | 0 | 8 | 5

BASELINE CHARACTERISTICS:
Population: For Part A, the Safety Analysis Set included all participants who received at least 1 dose of study drug in Part A.
Groups:
- Part A: Placebo: Participants weighing <50 kg drew equal volumes from two bottles of placebo oral solution to account for the daily dose assigned or participants weighing ≥50 kg received two placebo oral tablets, QD, during 12 weeks in Part A. Prucalopride matching placebo (oral solution or tablet) were dosed depending on the participant's BW at the randomization visit.
- Part A: Low Dose Prucalopride: Participants weighing <50 kg received 0.04 mg/kg of prucalopride oral solution (drew the required volume from one bottle of 0.4 mg/mL and one bottle of placebo oral solution), QD or participants weighing ≥50 kg received one 2 mg of prucalopride oral tablet and one placebo oral tablet, QD, during 12 weeks in Part A. Prucalopride (oral solution or tablet) were dosed depending on the participant's BW at the randomization visit.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Total
Number analyzed (Participants) | 56 | 60 | 59 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.4 (3.73) | 9.8 (4.00) | 9.8 (3.96) | 9.7 (3.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 28 | 91
  Male | 21 | 32 | 31 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 28 | 30 | 81
  Not Hispanic or Latino | 33 | 32 | 29 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 22 | 23 | 68
  White | 31 | 34 | 35 | 100
  More than one race | 0 | 2 | 0 | 2
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56 | 60 | 59 | 175
Weight [Mean (Standard Deviation); unit: kg] | 44.24 (25.318) | 47.24 (24.326) | 43.72 (23.793) | 45.10 (24.381)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 139.86 (23.563) | 142.57 (22.480) | 140.35 (24.554) | 140.96 (23.435)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = weight (kg)/[height (m)^2]
  kilograms per meter square (kg/m^2) | 20.76 (6.702) | 21.63 (6.461) | 20.44 (6.255) | 20.95 (6.454)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Average Number of Weekly Number of Spontaneous Bowel Movements (SBMs) at Week 12
Description: Spontaneous bowel movement was defined as a bowel movement that was not preceded within a period of 24 hours by the intake of rescue medication. The average change from baseline in number of SBMs per week derived from the (e-diary) data, in toilet-trained participants who were at least 3 years of age collected during the placebo-controlled part (Part A) was assessed.
Time Frame: Baseline, Week 12
Population: The Completers Analysis Set included all toilet-trained participants who were at least 3 years of age in the Modified Intent-to-treat Analysis Set (mITT) analysis set who had an average number of SBM available for all 12 weeks in the placebo-controlled part (Part A) of the study.
Measure: Mean (Standard Deviation); unit: SBMs per week
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride
Number analyzed (Participants) | 20 | 18 | 11
SBMs per week | 1.4 (1.90) | 1.9 (2.67) | 0.9 (1.44)

2. Primary Outcome: Parts A and B: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product that did not necessarily have a causal relationship with this treatment. A TEAE was defined as any event emerging or manifesting at or after the initiation of treatment with an investigational product (IP) or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. A serious adverse event (SAE) was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, is an important medical event.
Time Frame: From first dose of study drug up to Week 52
Population: For Part A, the Safety Analysis Set included all participants who received at least 1 dose of study drug in Part A. For Part B, the Safety Analysis Set included all participants who received at least 1 dose of study drug in Part B.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
Number analyzed (Participants) | 56 | 60 | 59 | 72 | 62
Participants
  TEAEs | 15 | 24 | 18 | 22 | 17
  TESAEs | 1 | 0 | 0 | 1 | 1

3. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters
Description: Laboratory parameters included blood chemistry, hematology, and urinalysis. Clinically significant laboratory parameters assessment was based on investigator interpretation. Number of participants with clinically significant changes in laboratory parameters (included hematology, blood chemistry, and urinalysis) were reported.
Time Frame: From first dose of study drug up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
Number analyzed (Participants) | 56 | 60 | 59 | 72 | 62
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Vital Sign Abnormalities
Description: Vital signs included measurement of pulse rate, systolic, and diastolic blood pressure. Clinically significant vital signs assessment was based on investigator interpretation. Number of participants with clinically significant changes in vital signs were reported.
Time Frame: From first dose of study drug up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
Number analyzed (Participants) | 56 | 60 | 59 | 72 | 62
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Parts A and B: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: ECG included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals parameters measurement. Clinically significant ECG assessment was based on investigator interpretation. Number of participants with clinically significant changes in ECG were reported.
Time Frame: From first dose of study drug up to Week 52
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
Number analyzed (Participants) | 56 | 60 | 59 | 72 | 62
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Part A: Change From Baseline in Participants' Weekly Stool Consistency Based on Bristol Stool Form Scale (BSFS) Score at Week 12 Categorized by Age
Description: The Bristol Stool Form Scale is a 7-score visual scale to measure stool consistency, 1- Separate hard lumps, hard to pass, 2- Sausage-shaped, but lumpy, 3- Like a sausage but with cracks on the surface, 4- Like a sausage or snake, smooth and soft, 5- Soft blobs with clear-cut edges, 6- Fluffy pieces with ragged edges, a mushy stool, 7- Watery, no solid pieces, entirely liquid. A score of 1 or 2 indicates constipation while a score of 6 or 7 indicates diarrhea. A better score (score of 3 and 4 represent ideal stools as they are easy to defecate while not containing excess liquid, 5 indicates average consistency but lack of dietary fiber) would trend toward the middle of the scale (3 to 5). Daily scores were summed to obtain a weekly score ranging from 7 to 49 with higher scores indicating diarrhea. Data for this outcome measure is reported per age group bifurcation.
Time Frame: Baseline, Week 12
Population: The mITT Analysis Set included all randomized participants who received at least 1 dose of the study drug in Part A. Overall number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride
Number analyzed (Participants) | 37 | 40 | 34
score on a scale
  Participants <8 Years: number analyzed (Participants) | 10 | 10 | 8
  Participants <8 Years | -0.1 (16.56) | 9.8 (12.75) | 7.1 (6.31)
  Participants ≥8 Years: number analyzed (Participants) | 27 | 30 | 26
  Participants ≥8 Years | 12.6 (16.77) | 13.1 (21.15) | 7.0 (10.44)

7. Secondary Outcome: Part A: Change From Baseline in Weekly Straining Score Based on a 3-point Likert Scale at Week 12
Description: Straining was assessed based on a 3-point Likert scale: (1=not at all, 2=a little, 3=a lot). A higher score indicates a lot of straining i.e., worsening of the condition. Daily scores were summed to obtain a weekly score ranging from 7 to 21 with higher scores indicating a lot of straining.
Time Frame: Baseline, Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride
Number analyzed (Participants) | 37 | 40 | 34
score on a scale | -5.7 (8.49) | -5.2 (5.92) | -7.6 (5.12)

8. Secondary Outcome: Part A: Percentage of Responders Based on Assessment of SBMs
Description: Spontaneous bowel movement was defined as a bowel movement that was not preceded within a period of 24 hours by the intake of rescue medication. Responder was defined as a participant having an increase of ≥1 SBM per week compared to Baseline and ≥3 SBMs per week for at least 9 out of the 12 weeks of placebo-controlled part (Part A), including 3 of the last 4 weeks. Percentages are rounded off to the nearest single decimal place.
Time Frame: Baseline through Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of responders
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride
Number analyzed (Participants) | 52 | 56 | 55
percentage of responders | 1.9 [0 to 0] | 3.6 [0 to 0] | 0 [0 to 0]

9. Secondary Outcome: Part A: Percentage of Participants With Fecal Incontinence at Week 12
Description: Fecal incontinence was defined as unintentional smear or liquid stool in the underwear that is not due to poor wiping. Fecal incontinence can only occur in toilet-trained participants. Non-retentive fecal incontinence is diagnosed (must include at least a 1-month history in a child with a developmental age older than 4 years for all the following): (i) defecation in places inappropriate to the sociocultural context, (ii) no evidence of fecal retention, and (iii) after appropriate evaluation, the fecal incontinence cannot be explained by another medical condition. Percentages are rounded off to the nearest single decimal place.
Time Frame: Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride
Number analyzed (Participants) | 31 | 33 | 30
percentage of participants | 12.9 [0 to 0] | 3.0 [0 to 0] | 16.7 [0 to 0]

10. Other Pre Specified Outcome: Part A: Pharmacokinetic (PK) Plasma Concentrations of Prucalopride
Time Frame: 1-3 hours post-dose at Baseline (Day 0), 14-26 hours post-dose at Weeks 4, 8 and 12
Population: The PK analysis set included all participants regardless of age in the safety analysis sets for whom at least 1 PK sample was evaluable. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride
Number analyzed (Participants) | 8 | 12
nanograms per milliliter (ng/mL)
  Baseline (Day 0), 1-3 hours: number analyzed (Participants) | 6 | 9
  Baseline (Day 0), 1-3 hours | 4.707 (3.4659) | 5.903 (4.0231)
  Week 4, 14-26 hours: number analyzed (Participants) | 7 | 8
  Week 4, 14-26 hours | 2.607 (0.7336) | 3.693 (2.0613)
  Week 8, 14-26 hours: number analyzed (Participants) | 6 | 6
  Week 8, 14-26 hours | 2.343 (1.8725) | 2.963 (2.0794)
  Week 12, 14-26 hours: number analyzed (Participants) | 6 | 6
  Week 12, 14-26 hours | 4.365 (3.6288) | 3.001 (4.5358)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 52
Description: For Part A, the Safety Analysis Set included all participants who received at least 1 dose of study drug in Part A. For Part B, the Safety Analysis Set included all participants who received at least 1 dose of study drug in Part B.
Arm/Group | Part A: Placebo | Part A: Low Dose Prucalopride | Part A: High Dose Prucalopride | Part B: Low Dose Prucalopride | Part B: High Dose Prucalopride
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/60 | 0/59 | 0/72 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/60 | 0/59 | 1/72 | 1/62
Other Adverse Events (participants affected / at risk) | 5/56 | 17/60 | 10/59 | 9/72 | 8/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=56) | Part A: Low Dose Prucalopride (N=60) | Part A: High Dose Prucalopride (N=59) | Part B: Low Dose Prucalopride (N=72) | Part B: High Dose Prucalopride (N=62)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=56) | Part A: Low Dose Prucalopride (N=60) | Part A: High Dose Prucalopride (N=59) | Part B: Low Dose Prucalopride (N=72) | Part B: High Dose Prucalopride (N=62)
Headache (Nervous system disorders) | 3 | 8 | 5 | 3 | 5
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 7 | 1
Vomiting (Gastrointestinal disorders) | 2 | 8 | 4 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT04759833/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT04759833/SAP_001.pdf